CLINICAL TRIAL: NCT05401604
Title: Probiotic Beer to Enhance Gut Health and Immune System Function
Acronym: PBEER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Mei Hui Liu, Co-Investigator, National University of Singapore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2021/00196
Record Dates: First submitted 2022-05-24; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Inflammation; Nutrition, Healthy
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: The experimental design used in this study is a randomised, controlled, within-subject cross-over design. Each individual will undergo a 2-week intervention each of moderate beer consumption and moderate probiotic beer consumption, with a 1-week period of washout in between. The total study duration will be 5 weeks.
Who Masked: Participant
Masking Description: Participants are blinded as to which beer (i.e. normal or probiotic) they are receiving for each intervention arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate probiotic beer consumption (Experimental): 1 can of 330ml (3.5-5% alcohol) probiotic beer. Ingredients: water, grains, raspberry puree, yeast, and lactic acid bacteria (Lactobacillus paracasei Lpc-37®, or Lactobacillus paracasei LAFTI®L26).
  Interventions: Dietary Supplement: Moderate probiotic beer consumption
- Moderate normal beer consumption (Placebo Comparator): 1 can of 330ml (3.5-5% alcohol) normal beer. Ingredients: water, grains, raspberry puree, and yeast.
  Interventions: Dietary Supplement: Moderate normal beer consumption

INTERVENTIONS:
Dietary Supplement: Moderate probiotic beer consumption — Consumption of one can of probiotic beer per day for 14 days. Blood and fecal samples will be collected at the start and end of the intervention to analyse for immunological biomarkers and gut microbiome.
  Arms: Moderate probiotic beer consumption
Dietary Supplement: Moderate normal beer consumption — Consumption of one can of normal beer per day for 14 days. Blood and fecal samples will be collected at the start and end of the intervention to analyse for immunological biomarkers and gut microbiome.
  Arms: Moderate normal beer consumption

SUMMARY:
This study investigates the immunological and gut microbiome effects of moderate probiotic beer consumption.

DETAILED DESCRIPTION:
Studies have shown that moderate alcohol consumption and probiotics have each shown immunomodulatory anti-inflammatory effects. However, to our knowledge, the effect of adding a probiotic strain to a beer drink, together with moderate alcohol consumption, on immunity and gut microbiome has yet to be studied. The probiotic beer used in this study taps on this unexplored research area and may potentially serve as a more healthful option to consumers than normal beer in the future, given the vast popularity of this beverage and probiotics.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent.
* 21 - 60 years of age (inclusive) at screening.
* Healthy male, as determined by medical history, physical examination and laboratory results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Race must be Chinese.
* Willing to consume 1 beer can per day for 14 days.
* Not on any regular medications (western/ traditional).
* No family history of alcoholism.

Exclusion Criteria:

* Female.
* A current smoker, have smoked, or is a user of tobacco products for the past 2 years.
* History or presence of current lipid and cardiovascular disorders, respiratory, hepatic, renal, gastrointestinal, endocrine, lipid disorder, haematological, malignancy or neurological disorders capable of significantly altering the performance of the biomarker panel; or of interfering with the interpretation of data.
* History of alcoholism, alcohol dependence, alcohol abuse, alcohol allergy and/or any other alcohol use disorders.
* History of Type 1/ Type 2 diabetes and use of anti-diabetic medications in the past.
* Regular use of medication that are known to have an effect on immune function.
* Regular use of aspirin.
* A naïve alcohol drinker.
* Persons with known or ongoing psychiatric disorders or drug abuse within 3 years.
* Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to first visit of the study.
* Treatment with any investigational drug, or biological agent within one (1) month of screening or plans to enter into an investigational drug/ biological agent study during the duration of this study.
* Significant change in weight (+/- 5%) during the past month.
* Antibiotic use in the past 2 months.

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Changes in inflammatory cytokine profile after moderate probiotic beer consumption. | 5 weeks
  Changes in inflammatory cytokine profile (IFNg, TNFa, IL-1b, IL-2, IL-4, IL-6, IL-10, IL-12) in blood samples of individuals after moderate probiotic beer consumption, in comparison to moderate normal beer consumption.
Changes in gut microbiome profile after moderate probiotic beer consumption. | 5 weeks
  Changes in gut microbiome profile from DNA sequencing in stool samples after moderate probiotic beer consumption, in comparison to moderate normal beer consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Hui Liu, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT05401604/Prot_SAP_000.pdf